CLINICAL TRIAL: NCT01555970
Title: Serotonin Reuptake Inhibitor Augmentation With N-Acetylcysteine in Resistant Obsessive-compulsive Disorder: a Double-blind, Randomized and Controlled Study
Brief Title: Efficacy Study of add-on Therapy With N-Acetylcysteine in Resistant Obsessive-compulsive Disorder
Acronym: NACTOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Roseli Shavitt, Psychiatrist, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NACTOC
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-compulsive disorder; Treatment; Glutamate; N-Acetylcysteine
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- NAC (Experimental): Patients allocated in this group will receive N-acetylcysteine 1200 mg (one 600 mg capsule twice a day) during the first week of the study. On day 8 this will increase to 4 capsules per day (2400 mg NAC; 2 capsules twice a day). Finally, on day 15 (after 1 week at 2400 mg) the dose will be increased to the target dose of 5 capsules per day (3000 mg; 2 capsules in the morning and 3 in the evening), at which dose it will be continued for the remainder of the study.
  Interventions: Drug: N-Acetylcysteine (NAC)
- Placebo (Placebo Comparator): Patients allocated in this group will receive one capsule of placebo twice a day during the first week of the study. On day 8 this will increase to 4 capsules per day (2 capsules twice a day). Finally, on day 15 the dose will be increased to the target dose of 5 capsules per day (2 capsules in the morning and 3 in the evening), at which dose it will be continued for the remainder of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine (NAC) — Week 1: 1200 mg (one 600 mg capsule twice a day) Week 2: 2400 mg (two 600 mg capsules twice a day) Weeks 3-16: 3000 mg (two 600 mg capsules in the morning and 3 in the evening)
  Arms: NAC
Drug: Placebo — Week 1: one capsule twice a day Week 2: two capsules twice a day Weeks 3-16: two capsules in the morning and 3 in the evening
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine if N-Acetylcysteine (NAC) has efficacy as an augmentation agent in the treatment of treatment-resistant obsessive-compulsive disorder (OCD). The investigators predict that NAC will reduce OCD symptoms after sixteen weeks of add-on treatment as measured by the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS).

DETAILED DESCRIPTION:
OCD is a debilitating psychiatric condition with a lifetime prevalence of 2-3%. It is characterized by recurrent, intrusive thoughts (obsessions) and/or repetitive, stereotyped behaviors (compulsions) that last for at least one hour per day and significantly interfere with an individual's normal level of functioning. Although cognitive behavioral therapy and pharmacotherapy with serotonin reuptake inhibitors (SRI) are effective treatments for many patients, a subset experience minimal relief from their symptoms with these standard treatments. When severe, OCD is completely incapacitating with devastating consequences for patients and their families. Augmentation strategies with antipsychotic medications can improve the effectiveness of SRI therapy but do no eliminate OCD symptoms (Saxena et al., 1996; McDougle et al., 1995) and are associated with adverse effects when used chronically; consequently, improved pharmacological treatments are needed. The clinical observation that few patients experience a complete response to SRI's or dopamine antagonists suggests that other neurochemical systems are involved in the pathophysiology of OCD.

The pathophysiologic hypothesis underlying this proposal is that the well-described hyperactivity of the cortico-striato-thalamic track in OCD reflects glutamatergic hyperactivity that is addressed only partially in some OCD patients by serotonin reuptake inhibitors treatment. It is thought that NAC modulates brain glutamate by stimulating the cysteine-glutamate antiporter located on glia, increasing extrasynaptic glutamate levels and thereby stimulating the feedback inhibition of synaptic glutamate release (Baker et al., 2003). In addition to attenuating synaptic glutamate release by feedback inhibition, NAC is also thought to enhance the clearance of glutamate from the synapse via its neuroprotective and growth factor promoting effects on glial cells. Its glutamatergic antagonistic properties may be effective in reducing the glutamatergic hyperactivity that is thought to contribute to the pathophysiology of OCD.

The proposed study is based on recent preclinical and neuroimaging studies that implicate glutamatergic hyperactivity in the pathogenesis of OCD (Carlsson et al., 2000). Neuroimaging studies have consistently identified increased blood flow, metabolism and brain activity in the orbitofrontal cortex, striatum, and thalamus of individuals with OCD (Baxter et al., 1987, 1988, 1992; Swedo et al., 1989; Sawle et al., 1991; Rubin et al., 1992, 1995; Adams et al., 1993; Perani et al., 1995; McGuire et al., 1994; Breiter et al., 1996; Rausch et al., 1996). Within these brain areas, glutamate and GABA driven pathways are thought to be responsible for balancing neural tone. The direct (glutamatergic) pathway is thought to modulate the initiation and sustainability of behavioral routines, while the indirect (GABAergic) pathway modulates the cessation of these behaviors. The leading explanatory model for OCD suggests that over activity in the direct pathway relative to the indirect pathway results in a disinhibited thalamus and the creation of a self-perpetuating circuit between the thalamus and the orbital cortex that drives OCD symptoms (Baxter 1992, Baxter et al., 1996). Clinical studies support this model. Compared to controls, treatment naïve OCD patients have significantly increased glutamatergic activity as measured by proton magnetic resonance spectroscopy (1H-MRS) (Rosenberg et al., 2000; Bolton et al., 2001). Moreover, treatment with an SRI was associated with a significant decline in caudate glutamate concentration in those individuals who responded to SRI treatment (Rosenberg et al., 2000; Bolton et al., 2001). These clinical findings are consistent with pharmacological studies demonstrating an SRI-induced inhibition of glutamate release (Maura et al, 1988; Zhang et al., 1997).

The investigators propose a double-blind, placebo controlled study to evaluate the tolerability and efficacy of N-Acetylcysteine in the augmentation of SRI therapy in resistant OCD. Four recent reports suggest that riluzole, an antiglutamatergic agent, possesses anti-depressant, anti-obsessional, and anti-anxiety properties (Coric et al., 2003, 2005; Zarate et al., 2004; Sanacora et al., 2004).

The rationale for exploring the efficacy of NAC in treatment resistant OCD stems from preliminary findings from the open label Riluzole study and represents an effort to explore other novel strategies for modulating brain glutamate in OCD.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signed informed consent prior to the performance of any study specific procedures
2. A DSM-IV primary diagnosis of OCD that has failed to clinically respond, as defined by a Y-BOCS score of greater than 16, to at least one first-line adequate treatments, like:

   * SRI
   * CBT
   * SRI + CBT
   * SRI + atypical antipsychotic
3. OCD symptoms at least of one year's duration and of least moderate severity on the Clinical Global Impression Scale (CGI).

Exclusion Criteria:

1. Psychiatric diagnosis of a primary psychotic disorder
2. Hepatitis or any liver disease
3. Patients who have had psychosurgery
4. Recent (<1 month) change in psychotropic medications
5. Presence of clinically significant somatic disease and/or medical problem that requires frequent changes in medication.
6. History of or current diagnosis of seizure disorder
7. Evidence of Substance Use Disorder (DSM-IV) within past 1 months or current illicit drug use.
8. Active Suicidal Ideation
9. Patients who have been previously exposed to N-acetylcysteine.
10. Women who are pregnant, lactating, or of childbearing potential (not sterile nor using reliable birth control).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale total score | 16 weeks
  Percent reduction of baseline Y-BOCS total score at weeks 16 or at withdrawal from the study

SECONDARY OUTCOMES:
Dimensional Yale-Brown Obsessive-Compulsive Scale score | 16 weeks
  The mean change in DYBOCS scores at week 16 or at withdrawal from the study
Clinical Global Impression Scale | 16 weeks
  Global Improvement score of the Clinical Global Impression Scale measured at week 16 or at withdrawal from the study
Beck Depression Inventory | 16 weeks
  The mean change in Beck Depression Inventory scores measured at week 16 or at withdrawal from the study
Beck Anxiety Inventory | 16 weeks
  The mean change in Beck Anxiety Inventory scores measured at week 16 or at withdrawal from the study

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Costa, MD, Principal Investigator — University of Sao Paulo; Roseli Shavitt, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Instituto de Psiquiatria do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Costa DLC, Diniz JB, Requena G, Joaquim MA, Pittenger C, Bloch MH, Miguel EC, Shavitt RG. Randomized, Double-Blind, Placebo-Controlled Trial of N-Acetylcysteine Augmentation for Treatment-Resistant Obsessive-Compulsive Disorder. J Clin Psychiatry. 2017 Jul;78(7):e766-e773. doi: 10.4088/JCP.16m11101. PMID 28617566